CLINICAL TRIAL: NCT00793494
Title: Randomized Controlled Trial of Probaclac Versus Placebo in Children Aged 8 to 18 Years With Irritable Bowel Syndrome
Brief Title: Efficacy of Probaclac in Irritable Bowel Syndrome in Children Aged 8 to 18 Years
Acronym: POPSII
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment impossible
Sponsor: St. Justine's Hospital (Other)
Collaborators: Nicar Inc. (Industry)
Responsible Party: Principal Investigator, Christophe Faure, MD, St. Justine's Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Probaclac-HSJ
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; Children; Pediatrics; Probiotics
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probaclac (Experimental): Administration of Bifidobacterium bifidum R0071, Bifidobacterium longum R0175, Lactobacillus helveticus R0052, Lactobacillus Delb. SSP bulgaricus R9001, Lactobacillus rhamnosus R0011, Lactococcus Lactis SSP. lactis R1058 et Streptococcus thermophilus (Probaclac™) b.i.d.
  Interventions: Other: Probaclac
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Probaclac — Bifidobacterium bifidum R0071, Bifidobacterium longum R0175, Lactobacillus helveticus R0052, Lactobacillus Delb. SSP bulgaricus R9001, Lactobacillus rhamnosus R0011, Lactococcus Lactis SSP. lactis R1058 et Streptococcus thermophilus (Probaclac™)
  Arms: Probaclac
Other: Placebo — Placebo composition matodextrin, gelatin, ascorbic acid, soya
  Arms: Placebo

SUMMARY:
The aim of this study is to determine the efficacy of the administration of Bifidobacterium bifidum R0071, Bifidobacterium longum R0175, Lactobacillus helveticus R0052, Lactobacillus Delb. SSP bulgaricus R9001, Lactobacillus rhamnosus R0011, Lactococcus Lactis SSP. lactis R1058 et Streptococcus thermophilus (Probaclac™) given twice a day for 4 weeks on digestive symptoms evaluated subjectively in children aged 8 to 18 years with irritable bowel syndrome versus placebo.

This study is a double-blind randomized controlled study. 84 children will included. After inclusion, a 15-day period of observation precedes the randomization at Day 0. Patients receive Probaclac or placebo for 4 weeks. At the end of the treatment period, patients are followed for a 2-week period of follow-up.

4 visits and 4 phone calls are planned during the study.

ELIGIBILITY:
Inclusion Criteria:

* Children 8 to 18 years
* Irritable bowel syndrome according to Rome III criteria

Exclusion Criteria:

* Not able to collaborate
* Known Digestive malformation
* History of digestive surgery (except hernia repair and appendectomy)
* History of known digestive disease (Crohn's, ulcerative colitis, esophagitis, peptic ulcer, celiac disease)
* Symptoms suggestive of organic disease (such as rectal bleeding, weight loss
* History of chronic extra-digestive disease
* Acute gastroenteritis in th e4 weeks prior to inclusion
* Central catheter, artificial cardiac valve, endocardiac prothesis
* Current Antidepressant treatment
* Patients taking a treatment for irritable bowel syndrome unable to cease their current treatment
* Patient taking regularly probiotics and natural products

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2009-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Subjective assessment of improvement of symptoms | 4 weeks

SECONDARY OUTCOMES:
Change in severity of symptoms (likert scale) | 4 weeks
Presence and intensity of pain episodes | 4 weeks
Presence or absence of urgency, incomplete evacuation, gas | 4 weeks
Number and consistance of the stools | 4 weeks
School and social absenteism | 4 weeks
Quality of Life | 4 weeks
Adverse Events | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Christophe M Faure, MD, Principal Investigator — Ste-Justine Hospital
Locations (1):
- Hôpital Sainte Justine, Montreal, Quebec, Canada

REFERENCES:
- See also: Related Info — http://www.christophefaure.org